CLINICAL TRIAL: NCT01024218
Title: An Open-label, Multicenter, Handling Test and Prospective Cross-over Study on Nurse/Health Assistants Preference Between NovoFine® Autocover™ and 8 mm NovoFine® Needle
Brief Title: Preference Study Between NovoFine® Autocover™ and a NovoFine® 8 mm Needle
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AUTOCOVER
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Healthcare Professionals; Delivery Systems
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: NovoFine® needle 8 mm
Device: autocover needle

SUMMARY:
This trial is conducted in Europe. The aim of this clinical trial is to assess the preference of 2 different needles used by nurses and health assistants. The trial consists of a handling test followed by a 12 week cross-over study.

ELIGIBILITY:
Inclusion Criteria:

* The participant must have been either a diabetes nurse or a diabetes health assistant with competence in subcutaneous injections of insulin for at least 4 weeks
* Participants must demonstrate proficiency with the injection device in the handling test prior to testing the NovoFine® Autocover™ Needle in patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2004-12-01 (Actual); Primary Completion 2005-04-26 (Actual); Study Completion 2005-04-26 (Actual)

PRIMARY OUTCOMES:
Device preference | after 12 weeks

SECONDARY OUTCOMES:
Comparison of the adverse device effects (occlusion/activation/locking problems/manufacturing defects)
Comparison of the frequency of adverse device effects
Comparison of the frequency of adverse events (needle stick injuries)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Copenhagen, Denmark

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com